CLINICAL TRIAL: NCT06684938
Title: Predictors of Outcome for Sacroiliac Joint Injection With Local Anaesthetic and Corticosteroids in Sacroiliac Joint Pain Patients
Brief Title: US Guided Sacroiliac Joint Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Sherine Elsherif, assistant professor, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0107462
Record Dates: First submitted 2024-10-15; First posted 2024-11-12 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2024-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- sacroiliac injection (Experimental): anaesthetic and steroid injection into the SIJ through US guidance
  Interventions: Drug: sacroiliac injection

INTERVENTIONS:
Drug: sacroiliac injection — sacroiliac injection with local anaesthetic and corticosteroids

SUMMARY:
Sacroiliac joint (SIJ) pain is one of the underappreciated causes of low back pain. Recent studies have reported excellent outcomes after Ultrasound (US) guided SIJ injection with local anesthetics and corticosteroids, but these studies are characterized by wide variability in selection criteria and patient characteristics; therefore, there is a need to determine whether any demographic or clinical variables can be used to predict US-guided SIJ injection outcomes.

DETAILED DESCRIPTION:
this study is testing the different predictors related to the patient that could affect his improvement by >50% after US guided SIJ injection with anaesthetic and steroids

ELIGIBILITY:
Inclusion Criteria:

* sacroiliac pain

Exclusion Criteria:

-

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
postinjection sacroiliac pain intensity | 3 months
  using Visual analogue scale for pain
postinjection disability questionnairre | 3 months
  using Modified Oswestry disability Questionnairre

CONTACTS AND LOCATIONS:
Overall Officials: SHERINE EL-SHERIF, Principal Investigator — Alexandria University
Locations (2):
- Egypt (2):
  - Sherine El-Sherif, Alexandria
  - Alexandria University, Alexandria